CLINICAL TRIAL: NCT02372422
Title: Use of Transvaginal Ultrasound Cervical Length Measurements in Twin Gestations
Brief Title: Transvaginal Ultrasound Cervical Length Measurements in Twin Gestations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William H. Barth, Jr., M.D., Col(ret), USAF, MC (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); Wright-Patterson Medical Center (Unknown)
Responsible Party: Sponsor-Investigator, William H. Barth, Jr., M.D., Col(ret), USAF, MC, William H. Barth, Jr., M.D., Col(ret), USAF, MC, 59th Medical Wing
Organization: 59th Medical Wing (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20020099H
Record Dates: First submitted 2015-02-15; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy
Keywords: Twins; Twin gestation; Preterm birth; Prevention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvaginal Cervical Length Group (Experimental): Clinicians managing the patients were aware of the transvaginal cervical length ultrasound measurements.
  Interventions: Other: Transvaginal ultrasound determination of cervical length
- Routine Care (Other): Clinicians managing the patients were not aware of any transvaginal cervical length ultrasound measurements.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Transvaginal ultrasound determination of cervical length — Transvaginal ultrasound was used to measure the length of the cervix from the internal to external os relying on a standard approach and clinicians caring for the patients were made aware of the results.
  Arms: Transvaginal Cervical Length Group
Other: Routine care — Routine prenatal care of twins. Digital exams were permitted, but transvaginal ultrasound assessment of cervical length was not.
  Arms: Routine Care

SUMMARY:
The purpose of this study is to determine if the use of routine transvaginal cervical length ultrasound can be used to prevent preterm deliveries in twin gestations.

DETAILED DESCRIPTION:
This is a randomized controlled trial to determine whether there is a difference in the rate of preterm birth among women with twin pregnancies whose clinicians are aware of transvaginal ultrasound cervical length measurements compared to those managed without this information. The study group had transvaginal cervical length ultrasound monthly from 16-28 weeks and were managed with a standard algorithm for activity restriction and cerclage depending on the cervical length. The control group had digital cervical exams and routine transvaginal cervical length ultrasound was not utilized. The primary outcome was the mean length of gestation. Secondary outcomes included percentage of deliveries < 35 weeks, maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy
* Gestational age < 20 weeks

Exclusion Criteria:

* History of incompetent cervix with plans to place a cerclage
* History of possible cervical incompetence with preexisting plans to monitor cervical length
* Prior preterm birth at < 28 weeks gestational age
* Plans to leave the area before delivery
* Known major fetal anomaly
* Known diagnosis of twin-twin transfusion syndrome
* Age < 18
* Monoamniotic twins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2002-10; Primary Completion 2006-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | Immediately at the time of delivery
  Gestational age reported as completed weeks of gestation

SECONDARY OUTCOMES:
Preterm birth at < 35 completed weeks of gestation | Immediately at the time of delivery
  The proportion of women delivering preterm at less than 35 completed weeks of gestation.
Number of days of maternal bed rest | Immediately at the time of delivery
  The number of days a woman was instructed to remain at bed rest or home rest before delivery
Number of maternal days in the hospital | Immediately at the time of delivery
  The number of antenatal hospital days not including the postpartum stay
Use of tocolytic medications | Immediately at the time of delivery
  Any use of tocolytic medications prior to delivery
Administration of steroids | Immediately at the time of delivery
  Any use of steroids for the promotion of fetal lung maturity
Birth weight | Immediately at the time of delivery
  Newborn birth weight
Length of stay in the neonatal intensive care unit | Newborns will be followed throughout their hospital stay for an anticipated average of 2 weeks
  Total days spent in the neonatal intensive care unit
Severe neonatal morbidity | Newborns will be followed throughout their hospital stay for an anticipated average of 2 weeks
  Composite outcome defined as one or more of the following: neonatal death, mechanical ventilation after 72 hours of life, chronic lung disease, grade 3 or 4 intraventricular hemorrhage or periventricular leukomalacia, necrotizing enterocolitis, stage 3 or higher retinopathy of prematurity, culture proven sepsis, or hemodynamic instability requiring pressor medications after 72 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Gordon, M.D., Principal Investigator — 59th Medical Wing